CLINICAL TRIAL: NCT05951400
Title: Progesterone Primed Ovarian Stimulation Protocol (PPOS) VS GnRH Antagonist Protocol in Patients With Expected High Ovarian Response Undergoing ICSI Cycles: a Prospective Randomized Controlled Trial
Brief Title: Progesterone Primed Ovarian Stimulation Versus GnRH Antagonist in With Expected High Ovarian Response Undergoing in Vitro Fertilization
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Sara Abdallah Mohamed Salem, Lecturer of Gynecology and obstetrics Faculty of medicine Beni-Suef University, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: duphaston in ICSI for PCO
Record Dates: First submitted 2023-06-04; First posted 2023-07-19 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: IVF; PCO
Keywords: Cetrorelix; Dydrogesterone; GnRh antagonist
MeSH Terms: interventions — Dydrogesterone; cetrorelix

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dydrogestrone (Experimental): For pituitary suppression, the patients will receive either Dydrogestrone (Duphaston 20 mg/d; Abbott Healthcare, USA) orally starting at day 2-3
  Interventions: Drug: Dydrogesterone Tablets
- GnRH antagonist (Active Comparator): For pituitary suppression, the patients will receive GnRH antagonist Cetrorelix (CETROTIDE 0.25Mg/d, Merck Serono, Germany) 0.25 mg/day subcutaneously from day 6 of induction until trigger day.
  Interventions: Drug: Cetrorelix

INTERVENTIONS:
Drug: Dydrogesterone Tablets — used for pituitary suppression in ICSI cycle
  Other Names: Duphaston
  Arms: Dydrogestrone
Drug: Cetrorelix — GnRH antagonist for pituitary suppression
  Other Names: cetrotide
  Arms: GnRH antagonist

SUMMARY:
To compare the effectiveness and safety of Progesterone Primed Ovarian Stimulation protocol (PPOS) using Dydrogestrone vs GnRH Antagonist Protocol in patients with expected high ovarian response undergoing ICSI cycle

DETAILED DESCRIPTION:
Each patient will be subjected to:

Full history taking. Systematic clinical examination to assess the general condition, body mass index (BMI) and local pelvic physical findings and AFC by trans-vaginal ultrasound on D2 to 3 of menstruation.

Routine labs as CBC, liver & kidney functions to exclude general disease as a contraindication for induction or pregnancy.

Blood sample will be obtained for assessment of basal serum levels of FSH, LH, E2 on days 2- 3 of the cycle. PRL, AMH and TSH Ovarian Stimulation The patients will begin injections of recombinant FSH (rFSH, Gonal-F; Merck-Serono, Italy) from day 2-3 of menstruation, with daily dose of 150-300 IU adjusted according to individual conditions on the basis of the antral follicle count (AFC),hormonal profile, age, body mass index (BMI), and previous ovarian response, according to the standard operating procedures of the center. .

For pituitary suppression, the patients will receive either Dydrogestrone (Duphaston 20 mg/d; Abbott Healthcare, USA) orally starting at day 2-3 or GnRH antagonist Cetrorelix (CETROTIDE 0.25Mg/d, Merck Serono, Germany) 0.25 mg/day subcutaneously from day 6 of induction until trigger day.

The serum LH, estradiol levels as well as number and size of follicles will be monitored every two days, starting from stimulation day 6 until the day of hCG injection. When most of dominant follicles reach diameter of 18-22 mm, the final oocyte maturation will be induced with 0.2 mg of Triptorelin (2 amp of Decapeptyl 0.1 mg, Ferring Pharmaceuticals, the Netherlands) (agonist trigger). Then, oocyte retrieval will be performed 34-36 h later with freezing of all embryos.

Frozen Embryo Transfer A maximum of 2 embryos will be transferred after endometrial preparation using Estradiol valerate(cycloprogenova 2mg tab Bayer Pharma AG, Germany) frome day 2 of cycle until endometrial thickness of 8 mm or more then adding progesterone 400 mg(Prontogest 400 IBSA pharmaceutical Italy) vaginal supp twice daily for 5 days and frozen embryo transfer will be on day 5 Transfer will be done by an expert using the same type of ET catheter under ultrasound guidance Adding progesterone 100 mg IM injection every other day if serum progesterone after 1st 4 doses of vag. Prog. is less than 9.2 ng/ml

An infant born alive after 22 weeks gestation was classified as a live birth. Clinical pregnancy is defined as the presence of at least 1 gestational sac on ultrasound at 6 weeks. Ongoing pregnancy is the presence of at least 1 fetus with heart pulsation on ultrasound beyond 10 weeks. Miscarriage rate was defined as the number of miscarriages before 24 weeks divided by the number of women with clinical pregnancy. Cancellation rate is defined as the number of patients with no viable embryos to transfer divided by the number of patients that started ovarian stimulation.

ELIGIBILITY:
Inclusion Criteria:

1. undergoing trial of ICSI.
2. BMI ≤ 30
3. AMH ≥3.5
4. AFC ≥ 20

Exclusion Criteria:

1. Any known contraindications to the approved fertility drugs.
2. Severe endometriosis.
3. Uterine malformations or abnormal uterine cavity.
4. Uncontrolled endocrinopathies:DM,hyperthyroidism, hypothyroidism
5. Severe male factor
6. History of recurrent ICSI failure or recurrent miscarriage

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-08-20 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
oocytes retrieved | 1 month of induction for ICSI trial
  Number of oocytes retrieved classified

SECONDARY OUTCOMES:
Duration of stimulation days. | 1 month
  number of days till giving trigger
chemical pregnancy rate | 1 month
  number of pregnancy test positive

CONTACTS AND LOCATIONS:
Overall Officials: Beni-Suef University, Principal Investigator — Faculty of Medicine Beni-Suef University
Locations (1):
- Beni-suef university Hospital, Banī Suwayf, Beni Suweif Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided